CLINICAL TRIAL: NCT05073614
Title: Evaluation of Immunohistochemical Expression of Heparanase in Helicobacter Pylori-Associated Chronic Gastritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maisa Hashem Mohammed, lecturer of pathology, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Soh-Med-21-09-43
Record Dates: First submitted 2021-09-19; First posted 2021-10-11 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Chronic Gastritis
Keywords: Heparanase; Chronic Gastritis; Helicobacter Pylori

STUDY DESIGN:
Intervention Model Description: patients with chronic gastritis will undergo upper endoscopy, punch biopsies will be obtained and tissue sections will be prepared from each specimen. sections will be stained by H&E to establish diagnosis of chronic gastritis. others will be stained by Giemsa staain to detect H.pylori, still others will be stained immunohistochemically by anti Heparanase antibody.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with chronic gastritis (Other): patients with symptomatic chronic gastritis will undergo upper endoscopy, gastric biopsies will be obtained to establish giagnosis of chronic gastritis, detection of h.pylori and assessment of heparanase expression.
  Interventions: Genetic: immunohistochemical detection of Heparanase in chronic gastritis

INTERVENTIONS:
Genetic: immunohistochemical detection of Heparanase in chronic gastritis — immunohistochemical detection of Heparanase in chronic gastritis specimens.

SUMMARY:
Treatment of H.pylori may not be achieved in many patients with chronic gastritis. Termination of the inflammatory respose produced by h.pylori may be useful in management of difficult cases. Heparanase is a pro-inflammatory mediator. Blocking of heparanase may relief the symptoms of chronic gastritis.

DETAILED DESCRIPTION:
Chronic gastritis (CG) is a very common disease. The incidence of CG is not accurately known. However, it is clear that the incidence of CG is increasing by advancing age. CG is divided into two main types; type A or immune and type B or non-immune gastritis. Both types of CG share the same histological features. However, type A is less common, usually affects the gastric fundus in a diffuse manner and separates the antrum. on the contrary; type B or non-immune CG, which is by far more common, inevitably develops in the antrum and progresses proximally. H. pylori-induced CG usually requires antibiotic therapy to eradicate the causative organism and subsequently terminate the inflammatory response and the symptoms of gastritis. However, eradication of H. pylori is difficult to be achieved in many patients. Previous studies established that there is a vicious circle between H. pylori-infected gastric epithelial cells and the gastric mucosal inflammatory cells. Heparanase (HPSE) is a mammalian ᵦ-endoglucoronidase. HPSE plays a critical role in multiple inflammatory processes by degrading and remodeling heparan sulfate polysaccharide chains in the extracellular matrix (ECM). This leads to release of multiple cytokines and chemokines which are located in the ECM. HPSE is a drug target, three inhibitors of this enzyme have been tested in early stage clinical trials. Many studies reported that the expression of HPSE is up-regulated in a variety of inflammatory conditions as ulcerative colitis, acute pancreatitis, acute vasculitis and sepsis. The aim of this work is to evaluate the role of heparanase (HPSE) in chronic gastritis (CG) by correlating the expression of HPSE to different histological features of CG as presence of H. pylori, chronic inflammatory infiltrate, gastric atrophy, intestinal metaplasia and neutrophil infiltrate (activity), to detect new treatment modalities in CG.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic chronic gastritis who underwent upper endoscopy.

Exclusion Criteria:

* patients with gastric carcinoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Correlation of Heparanase expression in chronic gastritis. | 6 months
  we will correlate the intensity and percentage of immunohistochemical expression of Heparanase to different parameters of chronic gastritis as severity of gastric atrophy, chronic inflammation, intensity of neutrophilic infiltrate and presence or absence of H. pylori.

CONTACTS AND LOCATIONS:
Locations (1):
- Maisa Hashem Mohammed, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No